CLINICAL TRIAL: NCT07208864
Title: Efficacy of an AI System in Training Endoscopists to Assess Gastric Intestinal Metaplasia Via the EGGIM Score: A Randomized Controlled Trial
Brief Title: Efficacy of an AI System in Training Endoscopists to Assess Gastric Intestinal Metaplasia Via the EGGIM Score
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2025SDU-QILU-4
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-05

CONDITIONS: Gastric Intestinal Metaplasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-assisted scoring first group (Experimental): Endoscopists will first evaluate the videos with the assistance of the AI system via EGGIM score, and after the washout period, the videos will be evaluated again without the assistance of the AI system.
  Interventions: Diagnostic Test: AI-assisted EGGIM scoring
- Conventional scoring first group (Active Comparator): Endoscopists will first evaluate the videos without the assistance of the AI system via EGGIM score, and after the washout period, the videos will be evaluated again with the assistance of the AI system.
  Interventions: Diagnostic Test: Conventional EGGIM scoring

INTERVENTIONS:
Diagnostic Test: AI-assisted EGGIM scoring — Endoscopists will evaluate the videos with the assistance of the AI system via EGGIM score.
  Arms: AI-assisted scoring first group
Diagnostic Test: Conventional EGGIM scoring — Endoscopists will evaluate the videos without the assistance of the AI system via EGGIM score.
  Arms: Conventional scoring first group

SUMMARY:
This prospective randomized controlled trial with a crossover design incorporated image-enhanced endoscopy (IEE) videos demonstrating complete standardized examinations of five standard gastric areas (antrum greater curvature, antrum lesser curvature, incisura, corpus lesser curvature, and corpus greater curvature). Endoscopists were stratified by experience level and randomly assigned to either the AI-assisted scoring first group, which performed EGGIM scoring with AI assistance in the initial phase followed by conventional scoring after a washout period, or the conventional scoring first group, which completed the assessments in reverse order. The study primarily evaluated the training efficacy of the EGGIM-AI system for improving endoscopists' EGGIM scoring performance by comparing diagnostic accuracy metrics including the area under the receiver operating characteristic curve (AUC), sensitivity, and specificity between groups at different study phases, with histopathological results serving as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

Endoscopists who have performed ≥50 image-enhanced endoscopy (IEE) procedures per year and demonstrated competency in performing standardized IEE.

Exclusion Criteria:

Endoscopists who participated in data acquisition or were unblinded to patients' identifiable information and clinical data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the EGGIM-AI system for improving endoscopists' EGGIM scoring performance | Through study completion, an average of 3 months
  Diagnostic accuracy metrics including the area under the receiver operating characteristic curve (AUC), sensitivity, and specificity between groups at different study phases, with histopathological results as the gold standard.

SECONDARY OUTCOMES:
Performance of EGGIM scoring by endoscopists with varying experience levels | Through study completion, an average of 3 months
  Differences in AUC, sensitivity, and specificity of EGGIM scores between experienced and inexperienced endoscopists within each group at different phases.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No